CLINICAL TRIAL: NCT04066881
Title: A Phase IIb Three-arm, Two-stage HIV Prophylactic Vaccine Trial With a Second Randomisation to Compare TAF/FTC to TDF/FTC as Pre-exposure Prophylaxis
Brief Title: A Combination Efficacy Study in Africa of Two DNA-MVA-Env Protein or DNA-Env Protein HIV-1 Vaccine Regimens With PrEP
Acronym: PrEPVacc
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MRC/UVRI and LSHTM Uganda Research Unit (Other)
Collaborators: Imperial College London (Other); University College, London (Other); International AIDS Vaccine Initiative (Network); EuroVacc Foundation (Other); Medical Research Council, South Africa (Other); National Institute for Medical Research, Tanzania (Other Government); Muhimbili University of Health and Allied Sciences (Other); Instituto Nacional de Saúde, Mozambique (Other Government); Ludwig-Maximilians - University of Munich (Other); King's College London (Other); Centre Hospitalier Universitaire Vaudois (Other); Karolinska Institutet (Other); CONRAD (Other); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RGPK190803
Record Dates: First submitted 2019-08-08; First posted 2019-08-26 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: HIV Infections
Keywords: HIV; Vaccine; Pre-exposure prophylaxis; Africa
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; emtricitabine tenofovir alafenamide

STUDY DESIGN:
Intervention Model Description: Group A: DNA-HIV-PT123/AIDSVAX B/E®/TDF/FTC (Truvada) once daily (wks 0-26) Group B: DNA-HIV-PT123 and CN54gp140+MPLA-L (wks 0,4), then MVA-CMDR and CN54gp140+MPLA-L/ TDF/FTC(Truvada) once daily (wks 0-26) Group C: Saline placebo (wks 0,4,24,48)/ TDF/FTC (Truvada) once daily (wks 0-26) Group D: DNA-HIV-PT123/AIDSVAX B/E®/ TAF/FTC (Descovy) once daily (wks 0-26) Group E: DNA-HIV-PT123 and CN54gp140+MPLA-L (wks 0,4), then MVA-CMDR and CN54gp140+MPLA-L/ TAF/FTC (Descovy) once daily (wks 0-26) Group F: Saline placebo (wks 0,4,24,48)/ TAF/FTC (Descovy) once daily (wks 0-26)
  Group G: Saline placebo (wks 0,4,24,48)/ TAF/FTC (Descovy) once daily (wks 0-26)
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The vaccine component of PrEPVacc is placebo-controlled. Study staff, participants, laboratory staff and clinical staff assessing safety outcomes will not know who has been allocated vaccine or placebo, but pharmacy staff will know. The committee assessing the efficacy endpoints will not see the allocation in the first instance. The IDMC and statistical staff preparing the closed reports for the IDMC will also know the allocation.
  Clinic staff will see the difference in volume between CN54gp140 in MPLA-L/matched placebo (0.4ml) and DNA-HIV-PT123/matched placebo (1ml) due to the position of the plunger, but they will not be able to differentiate between active and placebo.
  The randomisation to control PrEP: experimental PrEP is 1:1 and all study staff and participants will know the allocation after randomisation as this is open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Group A (Experimental): 278 participants will receive DNA-HIV-PT123 vaccine and AIDSVAX® B/E protein at weeks 0, 4, 24 and 48.
  1ml of DNA-HIV-PT123 will be injected into the deltoid muscle of the left upper arm
  1ml of AIDSVAX® B/E will be injected into the deltoid muscle of the right arm
  1 tab of Truvada (0-26 weeks)
  Interventions: Biological: Vaccine Group A: DNA-HIV-PT123 and AIDSVAX® B/E (weeks 0,4,24,48); Drug: Control PrEP:TDF/FTC once daily (weeks 0-26)
- Group B (Experimental): 278 participants will receive DNA-HIV-PT123 and CN54gp140+MPLA-L at weeks 0 and 4, then MVA and CN54gp140+MPLA-L at weeks 24 and 48
  1ml of DNA-HIV-PT123 will be injected into the deltoid muscle of the left upper arm
  1ml (1x108 pfu) of MVA will be injected into the deltoid muscle of the left upper arm
  0.4mL containing a mixture of 100mcg CN54gp140 and 5mcg MPLA-L will be injected into the deltoid muscle of the right upper arm
  1 tab of Truvada (0-26 weeks)
  Interventions: Biological: Vaccine Group B: DNA-HIV-PT123 and CN54gp140+MPLA-L (weeks 0,4), then MVA and CN54gp140+MPLA-L (weeks 24,48); Drug: Control PrEP:TDF/FTC once daily (weeks 0-26)
- Group C: (Placebo Comparator): 278 participants will receive Sodium Chloride 0.9% (Normal Saline) placebo at weeks 0,4,24, and 48
  The volume will be matched to the vaccine at 1ml for DNA, MVA and AIDSVAX® B/E, but 0.4ml for CN54gp140 in MPLA-L. Participants will be randomly divided in a 1:1 ratio to receive 1ml in each arm at the four timepoints or 1ml in the left arm and 0.4ml in the right arm at the four timepoints.
  1 tab of Truvada (0-26 weeks)
  Interventions: Biological: Vaccine Group C: Saline placebo (weeks 0,4,24,48); Drug: Control PrEP:TDF/FTC once daily (weeks 0-26)
- Group D (Active Comparator): 278 participants will receive DNA-HIV-PT123 vaccine and AIDSVAX® B/E protein at weeks 0, 4, 24 and 48.
  1ml of DNA-HIV-PT123 will be injected into the deltoid muscle of the left upper arm
  1ml of AIDSVAX® B/E will be injected into the deltoid muscle of the right arm
  1 tab of Descovy (0-26 weeks)
  Interventions: Biological: Vaccine Group A: DNA-HIV-PT123 and AIDSVAX® B/E (weeks 0,4,24,48); Drug: Experimental PrEP:TAF/FTC once daily (weeks 0-26)
- Group E (Experimental): 278 participants will receive DNA-HIV-PT123 and CN54gp140+MPLA-L at weeks 0 and 4, then MVA and CN54gp140+MPLA-L at weeks 24 and 48
  1ml of DNA-HIV-PT123 will be injected into the deltoid muscle of the left upper arm
  1ml (1x108 pfu) of MVA will be injected into the deltoid muscle of the left upper arm
  0.4mL containing a mixture of 100mcg CN54gp140 and 5mcg MPLA-L will be injected into the deltoid muscle of the right upper arm
  1 tab of Descovy (0-26 weeks)
  Interventions: Biological: Vaccine Group B: DNA-HIV-PT123 and CN54gp140+MPLA-L (weeks 0,4), then MVA and CN54gp140+MPLA-L (weeks 24,48); Drug: Experimental PrEP:TAF/FTC once daily (weeks 0-26)
- Group G (Placebo Comparator): 278 participants will receive Sodium Chloride 0.9% (Normal Saline) placebo at weeks 0,4,24, and 48
  The volume will be matched to the vaccine at 1ml for DNA, MVA and AIDSVAX® B/E, but 0.4ml for CN54gp140 in MPLA-L. Participants will be randomly divided in a 1:1 ratio to receive 1ml in each arm at the four timepoints or 1ml in the left arm and 0.4ml in the right arm at the four timepoints.
  1 tab of Descovy (0-26 weeks)
  Interventions: Biological: Vaccine Group C: Saline placebo (weeks 0,4,24,48); Drug: Experimental PrEP:TAF/FTC once daily (weeks 0-26)

INTERVENTIONS:
Biological: Vaccine Group A: DNA-HIV-PT123 and AIDSVAX® B/E (weeks 0,4,24,48) — 1. DNA-HIV-PT123 HIV vaccine includes three DNA plasmids that encode clade C ZM96 Gag, clade C ZM96 Env, and CN54 Pol-Nef.
  2. AIDSVAX® B/E is a bivalent HIV gp120 glycoprotein encompassing both subtype B (MN) and subtype E (A244) proteins that are adsorbed onto 600mcg of aluminum hydroxide gel suspension as adjuvant.
  Arms: Group A; Group D
Biological: Vaccine Group B: DNA-HIV-PT123 and CN54gp140+MPLA-L (weeks 0,4), then MVA and CN54gp140+MPLA-L (weeks 24,48) — 1. DNA-HIV-PT123 (see above)
  2. CN54gp140+MPLA-L. Recombinant CN54gp140 is a HIV-1 envelope protein from the clade C strain 97/CN/54 isolate, which comprises a sequence of 634 amino acids. MPLA is a non-toxic version of LipoPolySaccharide (LPS), which is isolated from the LPS lipid A region of Salmonella Minnesota R595 and retains the immune-stimulatory properties of LPS, but exhibits low toxicity.
  3. MVA-CMDR (Modified Vaccinia Ankara-Chiang Mai Double Recombinant) is a non-replicating, highly attenuated strain of Vaccina virus that has been genetically engineered to express the HIV-1 genes envgp160 CM235 Subtype E and gag and pol CM240 Subtype A (integrase-deleted and reverse transcriptase non-functional).
  Arms: Group B; Group E
Biological: Vaccine Group C: Saline placebo (weeks 0,4,24,48) — Sodium Chloride (NaCl) for injection, 0.9%
  Arms: Group C:; Group G
Drug: Control PrEP:TDF/FTC once daily (weeks 0-26) — Each tablet of Truvada contains 245mg of tenofovir disoproxil (TDF) and 200mg of emtricitabine (FTC), both of which are nucleot/side analogue HIV-1 reverse transcriptase inhibitors.
  Other Names: Truvada
  Arms: Group A; Group B; Group C:
Drug: Experimental PrEP:TAF/FTC once daily (weeks 0-26) — Each tablet of Descovy contains 25mg of tenofovir alfenamide (TAF) and 200mg of emtricitabine (FTC), both of which are nucleot/side analogue HIV-1 reverse transcriptase inhibitors.
  Other Names: Descovy
  Arms: Group D; Group E; Group G

SUMMARY:
This international, multi-centre, double-blind vaccine study is a three-arm prospective 1:1:1 randomisation comparing each of two experimental combination vaccine regimens i.e. DNA/AIDSVAX (weeks 0,4,24,48) and DNA/CN54gp140 (weeks 0,4) + MVA/CN54gp140 (weeks 24,48) with placebo control. There will be a concurrent open-label 1:1 randomisation to compare daily TAF/FTC (week 0-26) to daily TDF/FTC (weeks 0-26) as pre-exposure prophylaxis.

The study aims to randomise up to 1668 eligible adults (18-40 years) through collaborating clinical research centres in 4 countries (Mozambique; South Africa; Tanzania; and Uganda). Each participant will be followed for a minimum of 74 weeks after enrolment.

The trial is designed to detect a reduction in HIV incidence that has public health relevance sufficient to justify implementation of the combination vaccine regimen. In light of the high level of effectiveness demonstrated in the PrEP trials (up to 86% reduction in HIV), this trial is powered to detect a protective vaccine efficacy of 70% at the final analysis.

The PrEP component will determine whether the effectiveness of TAF/FTC is unacceptably lower than the effectiveness of TDF/FTC.

DETAILED DESCRIPTION:
This international, multi-centre, double-blind vaccine study will be a three-arm prospective 1:1:1 randomisation comparing each of two experimental combination vaccine regimens with placebo control.

Pre-screening for risk and HIV status will take place as part of a Registration Cohort which will precede and continue in parallel to the PrEPVacc trial enrolments. This will give HIV negative volunteers time to learn about the PrEPVacc trial and facilitate timely enrolment.

Clinical screening for the vaccine trial will take place during the 8 weeks prior to randomisation from local communities in Mozambique, South Africa, Tanzania and Uganda where the clinical research centres are located. Eligible participants who are HIV-uninfected adults aged 18-40 years at high risk of HIV infection will be enrolled at week 0 and randomised to one of three vaccine arms:

1. Vaccine group A: DNA-HIV-PT123 and AIDSVAX® B/E (weeks 0,4,24,48)
2. Vaccine group B: DNA-HIV-PT123 and CN54gp140 in MPLA-L (wks 0,4), then MVA-CMDR and CN54gp140 in MPLA-L (wks 24,48)
3. Vaccine group C: Saline Placebo (wks 0,4,24,48)

There will be a concurrent open-label 1:1 randomisation to one of two PrEP regimens:

1. Control PrEP: Daily TDF/FTC (week 0-26)
2. Experimental PrEP: Daily TAF/FTC (week 0-26)

Participants will be randomised at each clinical centre through web randomisation after entering the quantifiable eligibility criteria. Randomisation will be stratified by centre and by gender for vaccines and for PrEP. Clinic staff and participants will be blind to allocation of active or placebo vaccines, but the pharmacist preparing the vaccines will know. As the volume of gp140 in MPLA-L is 0.4ml and given at the same timepoints as products with a volume of 1ml, clinic staff will be able to identify participants allocated to the CN54gp140 in MPLA-L or matched placebo.

Clinic staff and participants will know which PrEP agent each participant is allocated to. Participants will continue to receive study PrEP through to week 26 after which access to PrEP will revert to local supply of generic drug.

The target accrual is around 1668 HIV uninfected adults, but this is an endpoint driven multi-arm, multi-stage (MAMS) trial design, and therefore the target may be adjusted following a recommendation from the IDMC. In addition, participants who do not complete the third immunisation will be replaced whilst this is feasible. Participants will be followed up for a minimum of 74 weeks after enrolment.

The primary efficacy outcome measure for the vaccine analysis is HIV acquisition by a participant who completed three immunisations and was HIV negative at week 26.

The primary efficacy outcome for the PrEP analysis is HIV acquisition at or before week 26 by a participant who was HIV negative at enrolment.

The primary safety outcome for both analyses is a clinical decision to discontinue the vaccine or PrEP regimen for an adverse event that is considered related to product.

This trial is designed to detect a reduction in HIV incidence that has public health relevance sufficient to justify implementation of the combination vaccine regimen. In light of the high level of effectiveness demonstrated in the PrEP trials (up to 86% reduction in HIV), this trial is powered to detect a protective vaccine efficacy of 70% at the final analysis.

The PrEP component of the trial aims to show the effectiveness of TAF/FTC is not unacceptably lower than the effectiveness of TDF/FTC, assessed from the observed lower confidence limit for the Averted Infections Ratio (AIR).

The Independent Data Monitoring Committee will review an interim analysis of vaccine efficacy in order to determine whether each active vaccine arm has demonstrated sufficient efficacy to warrant further investigation. This analysis will only consider new infections arising after the week 26 visit and only those in individuals who have completed the first three immunisations. The analysis will take place after approximately 7 of these infections have occurred in the placebo group. The investigators will not be informed of the timing of the interim analysis, unless there is a recommendation to modify the protocol.

The PrEP analysis will consider new infections up to the week 26 visit in individuals who were HIV negative at enrolment.

To enhance understanding of the trial results within their broader context, indepth interviews and group discussions with trial participants, as well as structured debriefs with study staff, will be conducted throughout the trial (week 0-74). These activities will examine risk and adherenvce behaviours, along with knowledge, attitudes and perceptions of participants, study staff and wider community.

ELIGIBILITY:
Inclusion criteria

1. HIV uninfected adults aged between 18 and 40 years old on the day of screening
2. Willing and able to provide informed consent prior to participation
3. Willing and able to comply with the visit schedule and provide blood, urine and other samples at the required time points
4. Home address accessible for visiting and intending to remain within the recruitment area for at least 82 weeks from screening
5. Likely to be at risk from exposure to HIV during follow up
6. Willing to undergo HIV testing, receive HIV test results and risk reduction counselling which includes promotion of PrEP and condoms
7. If female, of child-bearing age and not sterilised, willing to use a highly effective method of contraception from screening until 18 weeks after the last injection
8. If male and not sterilised, willing to avoid impregnating female partners from screening until 18 weeks after the last injection

Exclusion criteria

1. HIV infection or indeterminate HIV result at screening or enrolment
2. Hepatitis B surface antigen positive
3. If female, currently pregnant (evidence from positive serum or urine pregnancy test), or lactating
4. Participating in another biomedical research study or in receipt of a live vaccine within 30 days prior to randomisation
5. Participation in a previous HIV vaccine or HIV immunotherapy trial
6. Receiving blood products or immunoglobulins within 12 weeks of screening
7. Known hypersensitivity to any component of the vaccine formulations used in this trial or history of severe or multiple allergies to vaccines, drugs or pharmaceutical agents
8. Presence of a systemic disease at the time of randomisation or history of chronic illness that in the opinion of the investigator may compromise the participant's safety, preclude vaccination or compromise an immune response to vaccine
9. Abnormalities in routine laboratory parameters (Hb, creatinine, AST/ALT, alkaline phosphatase, total Bilirubin and glucose) of Grade 2 and above using the DAIDS toxicity table, version 2.1 July 2017 or estimated glomerular filtration rate less than 50ml/min

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1512 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Incident HIV infection | after week 26
  HIV acquisition by a participant who completed three immunisations and was HIV negative at week 26.
Incident HIV infection | week 0-26
  HIV acquisition at or before week 26 by a participant who was HIV negative at enrolment
A clinical decision to discontinue the vaccine regimen for an adverse event that is considered related to product | week 0-48
  A clinical decision to discontinue the vaccine regimen for an adverse event that is considered related to product
A clinical decision to discontinue PrEP regimen for an adverse event that is considered related to product | week 0-26
  A clinical decision to discontinue PrEP regimen for an adverse event that is considered related to product

SECONDARY OUTCOMES:
Grade 3 and worse solicited clinical and laboratory adverse events | week 0-74
  Grade 3 and worse solicited clinical and laboratory adverse events
Discontinuation or interruption of vaccine regimen | week 0-74
  A clinical decision to discontinue or interrupt the vaccine regimen for an adverse event that is considered related to product
Discontinuation or interruption of PrEP | week 0-26
  A clinical decision to discontinue or interrupt the PrEP regimen for an adverse event that is considered related to product
Grade 3 and worse solicited clinical and laboratory adverse events | within 7 days of receiving vaccine injection
  Grade 3 and worse solicited clinical and laboratory adverse events
Serious adverse events | week 0-74
  Serious adverse events
Other clinical and laboratory adverse events | week 0-74
  Other clinical and laboratory adverse events
Binding antibodies | week 0-74
  Binding antibodies to Cn54gp140 and AIDSVAX® B/E gp120
Resistance mutations to tenofovir and emtricitabine | week 0-74
  Genotypic resistance at HIV seroconversion, focussing on the mutations selected by tenofovir and emtricitabine (codons 65, 70, 184 in reverse transcriptase)
Number of PrEP pills missed | week 0-26
  Adherence to PrEP assessed by self-report
Tenofovir level in urine | week 0-26
  Adherence to PrEP assessed by results of point of care urine tests
Tenofovir level in red blood cells | week 0-26
  Adherence assessed by TFV DP levels measured on DBS in red blood cells
Number of PrEP Pills dispensed | week 0-26
  Adherence assessed by total number of PrEP pills dispensed

CONTACTS AND LOCATIONS:
Overall Officials: Pontiano Kaleebu, PhD, Principal Investigator — MRC/UVRI and LSHTM Uganda Resae; Sheena McCormack, MSc, Study Chair — MRC CTU at UCL; Jonathan Weber, PhD, Study Director — Imperial College London
Locations (1):
- MRC/UVRI and LSHTM Uganda Research Unit, Entebbe, Uganda

IPD SHARING:
Plan to Share IPD: Yes
The investigators will ensure that optimal use is made of the data generated in this trial through a controlled access approach to data sharing. Access will be controlled to ensure that there is a scientific rationale for the data, that no data are released that could compromise the ongoing trial, that the appropriate consent is in place, that an appropriate agreement is in place for secure transfer and storage, and that resources required to process data release are adequate.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The approved versions of the study protocol and global informed consent form will be in the public domain throughout.
  The Statistical Analysis Plan will be in the public domain prior to database lock.
  The clinical study report will be available a year after the last participant visit.
Access Criteria: The approved protocols and final version of the SAP will be in the public domain.
  The clinical study report will be available on request.

REFERENCES:
- [Derived] Ambikile JS, Tarimo EAM, Iseselo MK, Lukumay G, Munseri P, Bakari M, Lyamuya E, Aboud S, Kawuma R, Seeley J. The experience of trial participation disclosure among sex workers in a phase IIb HIV vaccine trial: A qualitative study in urban Tanzania. PLOS Glob Public Health. 2025 Nov 19;5(11):e0005511. doi: 10.1371/journal.pgph.0005511. eCollection 2025. PMID 41259346
- [Derived] Chimukuche RS, Shandu L, Zulu S, Khanyile P, Singh N, Gaffoor Z, Kawuma R, McCormack S, Seeley J; PrEPVacc Study Group. HIV risk perception, trust and PrEP adherence among participants in an HIV prevention trial: a qualitative longitudinal study, South Africa. BMJ Open. 2025 Apr 23;15(4):e086742. doi: 10.1136/bmjopen-2024-086742. PMID 40268488
- [Derived] Chimukuche RS, Kawuma R, Mahapa N, Mkhwanazi S, Singh N, Siva S, Ruzagira E, Seeley J; PrEPVacc Study Group. Examining oral pre-exposure prophylaxis (PrEP) literacy among participants in an HIV vaccine trial preparedness cohort study. BMC Health Serv Res. 2022 Nov 10;22(1):1336. doi: 10.1186/s12913-022-08730-8. PMID 36357877